CLINICAL TRIAL: NCT06964516
Title: A Prospective Randomized Controlled Study on Minimally Invasive Breast Effects Between the Modified Local Compression Bandaging Method and the Traditional Whole Breast Compression Bandaging Method
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2025-202-03
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Minimally Invasive Mammary Gland Vacuum-Assisted Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group using the whole-breast bandaging method (Active Comparator)
  Interventions: Procedure: The group using the whole-breast bandaging method
- The group using the local bandaging method (Experimental)
  Interventions: Procedure: The group using the local bandaging method

INTERVENTIONS:
Procedure: The group using the whole-breast bandaging method — Use 1 to 2 pieces of sterile loose gauze to knead into a gauze ball, press it on the residual cavity. Then, continue to use 5 to 8 pieces of loose gauze to stack gauze balls within a diameter of 5 cm around the wound for bandaging. Finally, apply compression bandaging with an elastic bra. The time for compression bandaging with the elastic bra is 24 hours.
  Arms: The group using the whole-breast bandaging method
Procedure: The group using the local bandaging method — Knead one or two pieces of loose gauze into a gauze ball to replace multiple gauze balls and place it in the residual cavity. Then, use elastic medical adhesive tape for local compression and sticking. Finally, place a pure cotton clean towel inside the elastic bra and wear the elastic bra for just one day.
  Arms: The group using the local bandaging method

SUMMARY:
I. Research Background Due to the relatively large trauma to the breast caused by traditional general anesthesia surgery, long recovery time, high incidence of postoperative complications, and patients' fear of general anesthesia surgery, the Mammotome minimally invasive rotary excision surgery has emerged. This minimally invasive breast surgery has very prominent advantages, mainly manifested as visualization, small incisions, and safety and reliability.

Currently, the commonly used bandaging method after minimally invasive breast surgery in clinical practice is the whole-breast compression bandaging method. One or two sterile loose gauze pieces are kneaded into a gauze ball and pressed on the residual cavity. Then, 5 to 8 loose gauze pieces are continuously stacked with the gauze ball within a 5 cm diameter around the wound for bandaging. Finally, an elastic bra is used for another day of compression bandaging. The elastic bra is a special compression elastic bandage for postoperative breast use to achieve auxiliary therapeutic effects such as clearing the cavity and protecting the surgical incision.

However, in the process of clinical practice, it has been found that this bandaging method brings great discomfort to patients. It is not only reflected in varying degrees of skin itching on the covered skin, and there are many cases of local red rashes. Moreover, it affects the patients' breathing. The vast majority of patients complain of pain and discomfort caused by the tight binding on the chest and back, feeling restless when sitting or lying down. At night, they can only sleep in a semi-sitting position and are largely unable to enter a deep sleep, seriously affecting the patients' daily activities and sleep conditions.

In order to improve the patients' experience and reduce their discomfort as much as possible, the medical and nursing joint team explored and improved the compression bandaging method after minimally invasive surgery and found that the local compression bandaging method is more comfortable. That is, one or two loose gauze pieces are kneaded into a gauze ball to replace multiple gauze balls and placed at the residual cavity. Then, elastic medical adhesive tape is used for local compression and sticking. Finally, a pure cotton clean towel is placed inside the elastic bra, and the elastic bra is worn for one day.

According to the results of a pre-experiment involving 50 cases, among the patients using the local compression bandaging method, there was no occurrence of wound hematoma, and their skin itching, chest and back pain, comfort level, and sleep conditions were all improved. In order to further compare the application effects of the whole-breast compression bandaging method and the local compression bandaging method, the research team of this study intends to conduct a comparative study of the two methods.

II. Research Objectives Research Objectives: Through a randomized controlled study, compare and study the curative effects of two different bandaging methods, namely the whole-breast bandaging method and the local bandaging method, during the perioperative period of minimally invasive breast surgery. Evaluate the impacts of the two bandaging methods on the wound healing situation after minimally invasive breast surgery, the incidence of hematoma, the patients' comfort level, and the incidence of patients' pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old.
2. The ultrasound report shows category 3 or category 4A.
3. Patients without allergy to medical adhesive tape.
4. Patients without hematopoietic system diseases such as bleeding tendency and coagulation dysfunction.
5. Willingly participate in the investigation and study.
6. No fever and no infection found during the admission physical examination.

Exclusion Criteria:

* 1. Patients with malignant breast tumors. 2. Patients with mental illnesses. 3. Patients who do not meet the indications for minimally invasive surgery according to the examination results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
The incidence of hematoma in patients: Use breast color Doppler ultrasound to check the wound healing condition and the presence of hematoma | At 2 weeks and 3 months after the operation respectively.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT06964516/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT06964516/ICF_001.pdf